CLINICAL TRIAL: NCT03915444
Title: A Phase II Trial of Nab-Paclitaxel Plus Cisplatin Plus Gemcitabine in Patients With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Nab-Paclitaxel + Cisplatin + Gemcitabine in Untreated Metastatic Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AX-CL-PANC-PI-13301
Record Dates: First submitted 2019-04-05; First posted 2019-04-16 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NabCG (Experimental): nab-paclitaxel 125mg/m2 cisplatin 25 mg/m2 gemcitabine 1000 mg/m2, all administered intravenously (IV) on Days 1 and 8 every 21 days
  Interventions: Drug: nab-Paclitaxel + Cisplatin + Gemcitabine

INTERVENTIONS:
Drug: nab-Paclitaxel + Cisplatin + Gemcitabine — Cisplatin 25mg/m2 in 500 mL of NS over 60 minute IV infusion on days 1 and 8 repeated every 21 days.
  Gemcitabine 1000mg/m2 in 500 mL* over 30 minute IV infusion on days 1 and 8 repeated every 21 days.
  Post cisplatin hydration: IV fluids up to 1000 mL (with additives as clinically indicated) IV given as infusion on days cisplatin is administered on days 1 and 8 repeated every 21 days.
  Other Names: NabCG

SUMMARY:
This is a phase II open-label study evaluating the efficacy and safety of nab-paclitaxel cisplatin, and gemcitabine in patients with metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This is a phase II open-label study evaluating the efficacy and safety of nab-paclitaxel cisplatin, and gemcitabine in patients with metastatic pancreatic ductal adenocarcinoma.

An individual cycle of therapy will be defined as Days 1 and 8 every 21 days. Multiple cycles may be administered until the patient is withdrawn from therapy.

Overall response rates as well as individual categories of response (CR, PR, SD, and PD) will be determined using RECIST 1.1 (Frese 2012). Time-to-event endpoints, including PFS and OS will be assessed using the Kaplan-Meier method (Kaplan 1958). Evaluation of stable disease at 9 weeks will also be assessed. Toxicity (adverse events) will be recorded using the NCI CTCAE, version 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age; male or female
2. Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma.
3. Capable of providing informed consent and complying with trial procedures.
4. Karnofsky Performance Status (KPS) of ≥ 70%.
5. Life expectancy ≥ 12 weeks.
6. Measurable tumor lesions according to RECIST 1.1 criteria.
7. < Grade 2 pre-existing peripheral neuropathy per NCI CTCAE, Version 5.0
8. Patient has acceptable coagulation status as indicated by an INR ≤1.5 x ULN. Patients on anticoagulation can be included at the discretion of the investigator.
9. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count ≥1,500/mm3
   * Platelet concentration ≥100,000/mm3 with no platelet transfusions within 7 days prior to laboratory sample
   * Hemoglobin > 9.0g/dL
   * Hematocrit level > 27%
   * Total bilirubin within 1.25 times institutional upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and AST < 10 × institutional ULN
   * Serum creatinine <1.5 mg/dl
10. Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

    1. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP therapy (including dose interruptions), and while on study medication or for a longer period if required by local regulations following the last dose of IP; and
    2. Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
11. Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following discontinuation from study treatment, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Patients must have received no previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatments in the neoadjuvant and/or adjuvant setting with gemcitabine and/or 5-FU based therapies or gemcitabine and/or 5FU administered as a radiation sensitizer are allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
2. Palliative surgery and/or radiation treatment less than 4 weeks prior to initiation of study treatment.
3. Exposure to any investigational agent within 4 weeks prior to initiation of study treatment.
4. Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
5. History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for ≥5 years.
6. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
7. History of HIV infection.
8. Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
9. Major surgery within 4 weeks prior to initiation of study treatment.
10. Any condition in the opinion of the principal investigator that might interfere with the patient's participation in the study or in the evaluation of the study results.
11. Any condition in the opinion of the principal investigator that is unstable and could jeopardize the patient's participation in the study.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
12- Month Overall Survival | 360 days
  Evaluate the 12-month OS rate in patients with metastatic PDA treated with nab-paclitaxel plus cisplatin plus gemcitabine

SECONDARY OUTCOMES:
Change in tumor markers | 63 days
  To determine the preliminary efficacy (Disease control rate of CR+ PR+SD X 9 weeks) of the combination of nanoparticle albumin- bound paclitaxel + cisplatin + gemcitabine (NABPLAGEM) in patients with stage IV metastatic pancreatic cancer.complete response rate( RECIST 1.1), disease control rate at 9 weeks, Change and rates of normalization in CA 19-9 (or Ca125 or CEA if not expressers of CA 19-9)
Quality of Life: MD Anderson Symptom Inventory (MDASI-GI) | 63 days
  Changes in patient's self-reported quality of life will be determined by administering the MD Anderson Symptom Inventory (MDASI-GI). This questionnaire asks about severity of symptoms using numbers (0 = not present to 10 = as bad as you can imagine).
Pain Control: Brief Pain Inventory (BPI) | 63 days
  Changes in patient's self-reported pain levels will be determined by administering the Brief Pain Inventory (BPI). This form asks about severity of pain using numbers (0 = not present to 10 = as bad as you can imagine).
Potential tumor biomarkers | 63 days
  Tumor biopsy testing will be completed to evaluate potential biomarkers in the tumor to evaluate various copy number variant signatures
Disease Response | 63 days
  Complete response rate as defined by CT scan using RECIST 1.1 criteria and CA 19-9 (or CA 125, or CEA if not expressers of CA 19-9) down to normal limits (from at least > 2X ULN).

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Jameson, ACNP-BC, Principal Investigator — HonorHealth Research Institute
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Miami, Miami, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No